CLINICAL TRIAL: NCT06120881
Title: Pilot Study of Precision Dosing of Metformin in Youth With Type 2 Diabetes (PRECISE_T2D)
Brief Title: Precision Dosing of Metformin in Youth With T2D
Acronym: PRECISE_T2D
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-39745; K23DK120932 (NIH)
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; metformin; pediatric
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): 1350mg metformin twice per day
  Interventions: Drug: Metformin
- Active Comparator (Active Comparator): 1000mg metformin twice per day
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Participants will receive either 2700mg of metformin/day (1350mg twice a day) or 2000mg of metformin/day (1000mg twice a day, standard of care). The study intervention will be blinded to the participants as they will receive the same number of pills (4 pills of the same size) regardless of whether they are in the intervention arm or control arm .

SUMMARY:
The purpose of this study to compare the typically prescribed dose of metformin (1000mg twice a day) with a higher dose of metformin (1350mg twice a day).

DETAILED DESCRIPTION:
Based on the investigators previous studies of young people who take metformin, the study team found that young people's bodies process metformin faster than older people and young people may need higher doses of metformin for the best treatment outcomes. The purpose of this study is to compare the typically prescribed dose of metformin (1000mg twice a day) with a higher dose of metformin (1350mg twice a day).

ELIGIBILITY:
Inclusion Criteria:

* Age 10-21 years
* Provider diagnosis of T2D
* Stable medication regimen for 2 weeks before screening visit (No addition or removal of medications and no more than 20% change in insulin dose)
* ≥ 1 month from T2D diagnosis
* Taking regular metformin (not extended-release formula)
* Ability to wear CGM for a total of 6 weeks while in the study.
* English or Spanish speakers.
* Willing to abide by recommendations and study procedures.
* Willing and able to sign the Informed Consent Form (ICF) and/or has a parent or guardian willing and able to sign the ICF.
* Participant and parent(s)/guardian(s) willingness to participate in all training sessions as directed by study staff. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Pancreatic autoantibody positivity (GAD-65, insulin, IA-2, ICA 512, Zn-T8).
* Known history of ongoing renal or hepatic disease.
* Known history of significant mental illness or developmental delay impacting the ability to complete study activities independently.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Higher Metformin Dose measured with the Acceptability of Intervention Measure (AIM) | Measured at 3 months
  The perception that a higher dose of Metformin is agreeable or satisfactory measured with the 4-item Acceptability of Intervention Measure (AIM). A 4-item measure of perceived intervention acceptability. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean. The greater the score, the better the acceptability.
Feasibility of Higher Metformin Dose measured with the Feasibility of Intervention Measure (FIM) | Measured at 3 months
  The extent to which a higher dose Metformin study can be successfully carried out measured with 4-item Feasibility of Intervention Measure (FIM). A 4-item instrument to assess perceived intervention feasibility. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean. The greater the score, the better the feasibility.

SECONDARY OUTCOMES:
Glycemic Change | Baseline (0) to 3 months
  Change in serum HbA1C at 3 months adjusted for the baseline value youth with T2D on higher dose of metformin compared to standard dose
Time in target glucose range | Baseline (0) to 3 months
  Time spent in target glucose range of 70 to 180 mg/dL
Time above high glucose range | Baseline (0) to 3 months
  Percent of readings and time >250 mg/dL
Time above glucose range | Baseline (0) to 3 months
  Percent of readings and time 181-250 mg/dL
Time in glucose range | Baseline (0) to 3 months
  Percent of readings and time 70-180 mg/dL
Time below glucose range | Baseline (0) to 3 months
  Percent of readings and time 54-69 mg/dL
Time below low glucose range | Baseline (0) to 3 months
  Percent of readings and time <54 mg/dl
Glucose management indicator | Baseline (0) to 3 months
  Continuous glucose monitoring (CGM) metric that indicates average blood glucose.
  Glucose Management Indicator (GMI) approximates the laboratory A1C level expected based on average glucose measured using CGM values. Average glucose is derived from 14 or more days of CGM readings.
Co-efficient of variation of glucose | Baseline (0) to 3 months
  CGM metric that measures variability in CGM values

CONTACTS AND LOCATIONS:
Overall Officials: Shylaja Srinivasan, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Pediatric Diabetes Clinic, Oakland, California
  - UCSF Benioff Children's Hospital San Francisco, Madison Clinic for Pediatric Diabetes, San Francisco, California

IPD SHARING:
Plan to Share IPD: No